CLINICAL TRIAL: NCT03264755
Title: Cortical Excitability and Role of rTMS in Nicotine Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Moheb, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEARORINUD
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-09

CONDITIONS: Nicotine Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cortical excitability in smokers (Active Comparator)
  Interventions: Device: Repetitive transcranial magnetic stimulation
- cortical excitability in nonsmokers (Active Comparator)
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation for cortical excitability in smokers and non smokers

SUMMARY:
Cortical excitability and role of repetitive transcranial magnetic stimulation in nicotine use disorder. Estimation of cortical excitability in heavy smoker patients and determination of role of repetitive transcranial magnetic stimulation for reducing nicotine craving.

DETAILED DESCRIPTION:
Nicotine is one of the main components of cigarettes and affects the central nervous system mainly via nicotinic acetylcholine receptors. It has further effects on neuromodulation by regulating the release of dopamine, serotonin, glutamate and adrenaline. In studies, it has been shown that nicotine improves attention and working memory in animals and humans, while nicotine withdrawal leads to reduced working and verbal memory capacity in otherwise healthy tobacco smokers. In schizophrenics and patients suffering from attention deficit hyperactivity disorder, nicotine improves cognitive performance. A likely basis of the nicotinic effects on cognitive functions is its effect on cortical excitability and activity. Here, neurophysiological studies mainly base on animal experiments and have shown in vitro that the nicotinic acetylcholine receptors elicit neuronal depolarisation by inducing transmembrane cationic inward currents (Calcium), thus being involved in induction and modulation of neuroplasticity and cortical excitability.

Repetitive transcranial magnetic stimulation: is a non-invasive brain stimulation technique that has shown positive results in the treatment of depression, schizophrenia, and more recently addiction. Repetitive transcranial magnetic stimulation uses alternating magnetic fields to induce electric currents in the cortical tissue. Low-frequency as one hertz repetitive transcranial magnetic stimulation is believed to inhibit neuronal firing in a localized area and is used to induce virtual brain lesions. High-frequency as more than three hertz repetitive transcranial magnetic stimulation is believed to be excitatory in nature and can result in neuronal depolarization under the stimulating coil. However, the effects of repetitive transcranial magnetic stimulation are not limited to the site of stimulation and can induce changes in distant interconnected sites of the brain, and consequently may influence subcortical regions.

ELIGIBILITY:
Inclusion Criteria:

1 )patients must be 18 to 50 years of age. 2) heavy smokers (daily cigarettes consumption of more than 20 pieces.)

Exclusion Criteria:

1. cardiac pacemaker.
2. metal implants in the head.
3. Renal diseases

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18 years
Enrollment: 60 (Estimated)
Dates: Start 2020-05-04 (Estimated); Primary Completion 2020-12-04 (Estimated); Study Completion 2020-12-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of cortical excitability between smoker and non smoker | 24 month
  Comparison of cortical excitability between smoker and non smoker :The primary motor cortex served as model, and cortical excitability was monitored via transcranial magnetic stimulation (TMS).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdelrahman AA, Noaman M, Fawzy M, Moheb A, Karim AA, Khedr EM. A double-blind randomized clinical trial of high frequency rTMS over the DLPFC on nicotine dependence, anxiety and depression. Sci Rep. 2021 Jan 15;11(1):1640. doi: 10.1038/s41598-020-80927-5. PMID 33452340